CLINICAL TRIAL: NCT05668481
Title: Improving Memory for Treatment for Patients Experiencing Mild Cognitive Impairment: Are Constructive or Non-constructive Memory Supports More Helpful?
Brief Title: Improving Patient Memory for Treatment for Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 2022-12-15881
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Memory Impairment; Sleep Disorder
Keywords: mild cognitive impairment; sleep and circadian functioning; improving treatment outcome
MeSH Terms: conditions — Memory Disorders; Sleep Wake Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive constructive memory supports in Session 1 OR to receive non-constructive memory supports in Session 1. In Session 2, participants will receive the type of memory support they did not receive in Session 1. In other words, if a participant received constructive memory support in Session 1, in Session 2 they will receive non-constructive memory support. And if a participant received non-constructive memory support in Session 1, in Session 2 they will receive constructive memory support. This cross-over design was adopted to increase the number of observations of the constructive and non-constructive memory support.
Who Masked: Participant
Masking Description: Participants will not be aware that they are receiving constructive memory support in one session and non-constructive memory support in the next session
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constructive memory support (Active Comparator): Participants will watch videos of a sleep expert delivering treatment components from the Transdiagnostic Sleep and Circadian Intervention (TranS-C). After each video, a team member will deliver constructive memory supports.
  Interventions: Behavioral: Transdiagnostic sleep and circadian intervention (TranS-C)
- Non-constructive memory support (Active Comparator): Participants will watch videos of a sleep expert delivering treatment components from the Transdiagnostic Sleep and Circadian Intervention (TranS-C). After each video, a team member will deliver non-constructive memory supports.
  Interventions: Behavioral: Transdiagnostic sleep and circadian intervention (TranS-C)

INTERVENTIONS:
Behavioral: Transdiagnostic sleep and circadian intervention (TranS-C) — TranS-C is a psychosocial treatment that helps people who have sleep and circadian problems to improve their sleep health.

SUMMARY:
The main empirical question to be addressed is: What types of memory support are most potent for patients who are experiencing a mild cognitive impairment (MCI) relative to non-MCI patients?

DETAILED DESCRIPTION:
People experiencing mild cognitive impairment (MCI) may benefit from adding memory support to treatment-as-usual. Adding memory support may be an innovative way to improve patient memory for treatment, adherence to treatment and outcome.

The key question is: What types of memory support are most potent for MCI patients relative to non-MCI patients?

The aim of the proposed research is to assess patient memory for treatment and the impact of adding memory support for people who are and are not experiencing MCI. The investigators will also compare the effectiveness of constructive vs. non-constructive memory supports for people who are experiencing MCI compared to people who are not experiencing MCI.

Hypotheses:

1. Recall of the content of treatment will be lower in the MCI group relative to the non-MCI group.
2. Constructive memory support will be more effective for the non-MCI group relative to the MCI group.
3. Non-constructive memory support will be more effective for the MCI group relative to the non-MCI group.

The outcomes are: (1) patient memory for the content of treatment session and (2) the number and accuracy of thoughts and applications of the therapy points delivered. The investigators will also collect ratings of the acceptability of the treatment and the memory supports that are delivered.

This dataset will also be used to better understand the sleep and circadian challenges that people with and without MCI report via the SCID for sleep disorders and the PROMIS scales.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 60 years and older will be recruited.
2. Fluent in English.
3. Experiencing some difficulties relating to sleep and circadian functioning and (d) a score of 19-25 on the Montreal Cognitive Assessment (for the MCI group) and score 26-30 on the Montreal Cognitive Assessment (for the non-MCI group) (e) Have a computer to use and an internet connection and (f) be able to attend sessions weekly and on the same day each week.

Exclusion criteria:

1. Presence of an active and progressive mental or physical illness or neurological degenerative disease;
2. Night shift work >2 nights per week in the past 3 months;
3. Not able and willing to participate in and/or complete the assessments and participate in the treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Number of items recalled on the free recall task to assess outcome for constructive memory support | Delivered two times: At the session in which constructive memory supports were used (baseline) and 1 week later.
  Assesses patient memory for treatment
Number of items recalled on the free recall task to assess outcome for non-constructive memory support | Delivered two times: At the end of the session in which non-constructive memory supports were used (baseline) and 1 week later.
  Assesses patient memory for treatment
Number and accuracy of thoughts about the material covered in the prior treatment session in which constructive memory supports were delivered | Delivered once: At the beginning of the session held 1 week after the delivery of the constructive memory supports
  To assess if the participant thought about the therapy session and if the thoughts accurately reflected the prior treatment session
Number and accuracy of thoughts about the material covered in the prior treatment session in which non-constructive memory supports were delivered | Delivered once: At the beginning of the session held 1 week after the delivery of the non-constructive memory supports
  To assess if the participant thought about the therapy session and if the thoughts accurately reflected the prior treatment session
Number and accuracy of applications of the material covered in the prior treatment session in which constructive memory supports were delivered | Delivered once: At the beginning of the session held 1 week after the delivery of the constructive memory supports
  To assess if the participant applied the material covered in the therapy session and if the participant accurately applied the material prior treatment session
Number and accuracy of applications of the material covered in the prior treatment session in which non-constructive memory supports were delivered | Delivered once: At the beginning of the session held 1 week after the delivery of the non-constructive memory supports
  To assess if the participant applied the material covered in the therapy session and if the participant accurately applied the material prior treatment session

SECONDARY OUTCOMES:
Acceptability of constructive memory support | One time point: At the end of the treatment session in which constructive memory support was delivered
  Participants will be asked to rate the "How acceptable were the memory supports we asked you through this session?" The participant will then provide a rating from "1" Not at all acceptable to "9" Very acceptable.

OTHER OUTCOMES:
PROMIS-Sleep Disturbance | At baseline
  Assesses perceived functional impairments related to sleep problems using a self-report questionnaire. The minimum value is 8. The maximum value is 40. Higher scores mean more sleep disturbance (worse outcome).
PROMIS-Sleep-related impairment | At baseline
  Assesses perceived functional impairments related to sleep problems in a self-report questionnaire. The minimum value is 16. The maximum value is 80. Higher scores mean more sleep related problems (worse outcome).
British Columbia Cognitive Complaints Inventory | At baseline
  Assessed perceived cognitive difficulties, scale consists of 6 items. Scores can range from 0-18 with higher scores indicating higher levels of perceived cognitive difficulties
Cognitive Failures Questionnaire | At baseline
  Used to assess the frequency with which people experienced cognitive failures. Scores range from 0-100, with higher scores indicating higher levels of cognitive failures.
Montreal Cognitive Assessment | At baseline
  An assessment of cognitive functioning
Structured Clinical Interview for Sleep Disorders - revised | At baseline
  An assessment of the sleep and circadian problems experienced by the participant
Learning behavior exhibited by the patient | Two time points: During the treatment session that constructive memory support was delivered and during the treatment session that non-constructive memory support was delivered
  Coded from video tapes of the two treatment sessions in which the support was delivered
Signs of patient understanding the memory support items | Two time points: During the treatment session that constructive memory support was delivered and during the treatment session that non-constructive memory support was delivered
  Coded from video tapes of the two treatment sessions in which the support was delivered

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States